CLINICAL TRIAL: NCT01242280
Title: Esophageal Stent is More Effective Than Tamponade Controlling Refractory Esophageal Variceal Bleeding: a Randomized Controlled Trial
Brief Title: Self-expandable Esophageal Stent Versus Balloon Tamponade in Refractory Esophageal Variceal Bleeding.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); Hospital Universitario Ramon y Cajal (Other); Puerta de Hierro University Hospital (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario Central de Asturias (Other)
Responsible Party: Principal Investigator, Angels Escorsell, Consultant. Liver Unit, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PE08001
Record Dates: First submitted 2010-08-04; First posted 2010-11-17 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Esophageal Varices; Bleeding; Cirrhosis
Keywords: Acute variceal bleeding; Massive bleeding; Liver Cirrhosis; Esophageal tamponade; Esophageal stent
MeSH Terms: conditions — Esophageal and Gastric Varices; Hemorrhage; Fibrosis; Liver Cirrhosis | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-expandable esophageal stent (Active Comparator): The patient will receive a self-expandable esophageal stent (SX-Ella-Danis) without endoscopical guidance but under slight sedation. An immediate X-ray will be done to assess the correct placement of the stent.
  After a maximum of 7 days, the stent will be removed by using the specifically designed devices.
  Interventions: Device: Stent
- Sengstaken-Blakemore tube (Active Comparator): The esophageal tamponade will be done as described elsewhere. The gastric content will be checked hourly and the correct placement of the tube will be checked by an immediate X-ray. The esophageal balloon will be inflated a maximum of 24 hours.
  Interventions: Device: Tamponade

INTERVENTIONS:
Device: Stent — Self-expandable esophageal stent (SX-Danis, Czesc Republic).
  Arms: Self-expandable esophageal stent
Device: Tamponade — Sengstaken-Blakemore tube
  Arms: Sengstaken-Blakemore tube

SUMMARY:
In the last years, important advances have been done in the treatment and prevention of esophageal variceal bleeding. Experts agree that the combination of pharmacological and endoscopic therapy should be the first line therapy in the acute bleeding episode; whereas TIPS (transjugular intrahepatic portosystemic shunt) is considered a rescue therapy. Nevertheless, some patients would require different therapies to act as a "bridge" until definitive therapy can be instituted. Balloon tamponade (using the Sengstaken tube) represents, up to now, the most widely used temporary "bridge" to TIPS. However, balloon tamponade is associated with a high incidence of serious adverse events. Recently, the use of self-expanding metal stents have been introduced in the treatment of acute variceal bleeding showing a very high hemostatic efficacy with no adverse events. The present study is directed to compare the efficacy free of adverse events and mortality of self-expanding metal stents vs balloon tamponade in patients with variceal bleeding refractory to medical and endoscopic therapy.

DETAILED DESCRIPTION:
BACKGROUND Acute variceal bleeding (AVB) carries a 20% death rate during the acute episode and nearly 50% related-mortality during the first year after the episode. (1). Prognostic factors of AVB include: the severity of bleeding, the degree of liver failure and the development of complications other than bleeding.

Therefore, AVB therapy must: achieve primary hemostasis and prevent and treat both hypovolemia and related complications. After hemodynamic stabilization, upper endoscopy should be done to confirm the diagnosis and start specific therapy, that is to say: 1/ vasoactive drugs (terlipressin or somatostatin); and 2/ endoscopic therapy (variceal banding ligation). These two combined therapies achieve control of AVB in 80% of the cases (2). Nevertheless, in the remaining 20%, the AVB is not controlled requiring balloon-tamponade as a bridge to definitive hemostatic therapies such as TIPS or surgical shunts(3). The Sengstaken-Blakemore tube is the most widely used balloon tamponade. In experienced hands it provides bleeding control rates up to 90%. It should only be used by skilled staff in intensive care facilities because fatal complications may arise in more than 20% of cases. The main complications are: aspiration pneumonia, esophageal rupture, asphyxia due to balloon migration, esophageal ulcers, tongue or nose or lips necrosis, arrythmia and chest pain. These complications are time-related, therefore, balloon tamponade never must remain inflated more than 24h.

Recently, a self-expandable esophageal stent has been introduced as an alternative to esophageal balloon tamponade in AVB (4). Twenty patients with AVB not controlled with combined endoscopic and pharmacological therapy were retrospectively included in the study. The patients received a self-expandable metal esophageal stent (SX-Ella-Danis, Czesc Republic). The stent was placed without complications in all cases achieving a 100% success in the control of AVB. Two to 14 days after, the stents were retired. The authors observed no case of severe stent-related complications and no rebleeding episodes (4).

These data suggest that self-expandable esophageal stent could represent a safe and effective option to temporary treat patients with AVB refractory to medical and endoscopic therapy. In addition, and theoretically, esophageal stent could be associated with a lower incidence of adverse events than balloon tamponade.

EXPECTED RESULTS

The initial hypothesis are:

* The use of esophageal stents in AVB refractory to medical and endoscopic therapy is associated with a higher efficacy in absence of adverse events than balloon tamponade using the Sengstaken-Blakemore tube.
* The two hemostatic methods are correctly positioned in more than 90-95% of the cases.
* Patient's tolerability (absence of chest pain, dysphagia or food intolerance) increases with the use of esophageal stents.
* The applicability of definitive hemostatic therapy, such as TIPS or combined pharmacological and endoscopic eradicative therapy or surgical shunts, is higher with the use of esophageal stents that with that of the Sengstaken tube.

ENDPOINTS

Primary endpoint:

The primary endpoint combines absence of bleeding + absence of severe adverse events probably related to the study devices + survival during the first 15 days after inclusion in the study or at hospital discharge.

Patients to compare are those with liver cirrhosis and AVB not controlled with combined pharmacological and endoscopic therapy (see definitions). Those patients will be randomized to receive a self-expandable esophageal stent (SX-Ella-Danis) or balloon tamponade with a Sengstaken-Blakemore tube.

Secondary endpoints:

* Absence of bleeding at day 15th, 42nd and at 6 months from inclusion.
* Survival at day 15th, 42nd and at 6 months from inclusion.
* Transfusional requirements (packed red cells, platelets and fresh frozen plasma).
* Individual adverse events.
* Analgesia and sedation requirements.
* Hospital stay.
* Applicability of definitive hemostatic therapy.
* Use of hospital resources (TIPS, derivative surgery or additional endoscopic therapy).

SAMPLE SIZE

The studies used to calculate the sample size are shown as references 7 to 22. None of these studies has considered a combined end-point such as in the current study.

As shown, the incidence of adverse events varied over time, the highest incidence being observed in the most recent studies. In summary, we have considered that 55% of the patients receiving esophageal balloon tamponade will achieve our primary end-point. To increase this figure to 90% in the group receiving esophageal prothesis, with an 0.05 alpha error and a 0.20 beta error, the study must include 46 patients (23 per arm).

STATISTICAL ANALYSIS

The results will be analyzed on an intention-to-treat basis. The data will be compared by using Student t test or Chi-squared as needed. Probability and survival curves will be constructed by using the Kaplan-Meier method and compared by the Mantel-Cox test. Logistic regression will be used to identify independent predictors of survival.

An interim analysis was planned after the inclusion of 28 patients (60% of the overall size). The study will be finished if the interim analysis shows significant statistical differences (p<0.02) or futility (lack of differences).

ELIGIBILITY:
Inclusion Criteria:

The study will include all patients with cirrhosis admitted to the hospital because an acute esophageal variceal bleeding defined according to Baveno II criteria (5) and who will achieve the following criteria:

* Failure to control bleeding despite pharmacological (somatostatin 3 or 6 mg/12h iv or terlipressin, 2mg/4h iv) AND endoscopic therapy (esophageal banding ligation preferably or sclerotherapy). Failure to control bleeding was defined, according to Baveno IV criteria (6), as evidence of continuous digestive bleeding and any of the following:

  * Hematemesis (or naso-gastric aspirate > 100 ml of fresh blood) > 2h after the start of combined pharmacological and endoscopic therapy.
  * Decrease in hemoglobin values > 3g vs previous values (without blood transfusion).
* Massive bleeding. Acute variceal bleeding uncontrolled despite pharmacological therapy started at any moment, with no need of previous endoscopic therapy. Uncontrolled bleeding is defined as an upper digestive bleeding in which no hemodynamic stability (systolic arterial pressure > 70 mmHg and heart rate < 100 bpm) could be achieved.

Exclusion Criteria:

* Age < 18 years.
* Esophageal rupture.
* Esophageal, gastric or upper respiratory tract tumor.
* Esophageal stenosis.
* Recent esophageal surgery.
* Previous esophageal tamponade to treat the index bleed.
* Big hiatal hernia precluding the correct placement of the esophageal devices.
* Known hepatocellular carcinoma surpassing Milan criteria.
* Terminal disease.
* No written consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Combined: bleeding + absence of severe adverse events + survival | 15 days
  The primary endpoint combines absence of bleeding + absence of severe adverse events probably related to the study devices + survival during the first 15 days after inclusion in the study or at hospital discharge.
  Patients to compare are those with liver cirrhosis and acute variceal bleeding (AVB) not controlled with combined pharmacological and endoscopic therapy (see definitions). Those patients will be randomized to receive a self-expandable esophageal stent (SX-Ella-Danis) or balloon tamponade with a Sengstaken-Blakemore tube.

SECONDARY OUTCOMES:
Bleeding | 6 months
  • Absence of bleeding at day 15th, 42nd and at 6 months from inclusion.
Survival | 6 months
  • Survival at day 15th, 42nd and at 6 months from inclusion.
Transfusional requirements | 15 days
  • Transfusional requirements (packed red cells, platelets and fresh frozen plasma).
Adverse events | 15 days
  • Individual adverse events.
Analgesia and sedation requirements | 15 days
  • Analgesia and sedation requirements
Hospital stay | 6 months
  • Hospital stay
Applicability of definitive hemostatic therapy. | 15 days
  • Applicability of definitive hemostatic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Angels Escorsell, MD, Principal Investigator — Liver Unit. Hospital Clínic
Locations (1):
- Hospital Clinic, Barcelona, Spain

REFERENCES:
- [Derived] Escorsell A, Pavel O, Cardenas A, Morillas R, Llop E, Villanueva C, Garcia-Pagan JC, Bosch J; Variceal Bleeding Study Group. Esophageal balloon tamponade versus esophageal stent in controlling acute refractory variceal bleeding: A multicenter randomized, controlled trial. Hepatology. 2016 Jun;63(6):1957-67. doi: 10.1002/hep.28360. Epub 2016 Jan 14. PMID 26600191